CLINICAL TRIAL: NCT01980056
Title: A Phase 1/2, Open-label, Dose Escalation Clinical Study of the Safety and Clinical Activity of Vosaroxin in Patients With Intermediate 2 or High-risk Myelodysplastic Syndrome (MDS) After Failure of Hypomethylating Agent-based Therapy
Brief Title: Vosaroxin for Intermediate 2 or High-risk MDS After Failure With Hypomethylating Agent-based Therapy
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Weill Medical College of Cornell University (Other)
Collaborators: Sunesis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: 1305013919; IST/VOS/MDS (Other: Weill Cornell Medical College)
Record Dates: First submitted 2013-11-01; First posted 2013-11-08 (Estimated); Results first posted 2018-12-28 (Actual); Last update posted 2019-02-19 (Actual); Status verified 2019-01

CONDITIONS: Myelodysplastic Syndrome
Keywords: INT-2 or high-risk MDS
MeSH Terms: conditions — Myelodysplastic Syndromes | interventions — vosaroxin

STUDY DESIGN:
Intervention Model Description: Dose level 1: Vosaroxin 50 mg/m^2 IV on Days 1 and 4 of 28 day cycle Dose level 2: Vosaroxin 72 mg/m^2 IV on Days 1 and 4 of 28 day cycle Dose level 3: Vosaroxin 50 mg/m^2 IV on Days 1, 4, 8 and 11 of 28 day cycle
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Vosaroxin: All Patients (Experimental): All patients will receive vosaroxin according to the dose cohort in which they are enrolled.
  Interventions: Drug: Vosaroxin

INTERVENTIONS:
Drug: Vosaroxin — Dose level 1: Vosaroxin 50 mg^m2 IV on Days 1 and 4 of 28 day cycle Dose level 2: Vosaroxin 72 mg^m2 IV on Days 1 and 4 of 28 day cycle Dose level 3: Vosaroxin 50 mg^m2 IV on Days 1, 4, 8 and 11 of 28 day cycle
  Other Names: Qinprezo

SUMMARY:
Study WCMC IST/VOS/MDS evaluates the safety and tolerability of escalating doses of vosaroxin in adult patients with pathologically confirmed Myelodysplastic Syndrome, or MDS, (< 20% blasts in bone marrow, peripheral blood, or both) by World Health Organization (WHO) classification with an intermediate 2 (INT-2) or high-risk score (ie, ≥ 1.5) as assessed by the International Scoring System (IPSS) after failure of hypomethylating agent-based therapy. Based on 3 completed studies and xenograft models, Vosaroxin is hypothesized to be safe and will effective in this patient population.

DETAILED DESCRIPTION:
This is a phase 1-2, dose escalation study of the safety and clinical activity of vosaroxin in subjects with INT-2 or high risk MDS who have failed prior hypomethylating agent based therapy. The study will utilize a standard 3+3 design to estimate the MTD [maximum tolerated dose] for vosaroxin administered to subjects with MDS. MTD will be defined as the highest dose level at which no more than 33% of the subjects observed at a given dose level experience a DLT [dose limiting toxicity]. Subjects will be assessed for safety and DLT in the first cycle of vosaroxin. Subjects will be enrolled into the study in cohorts of 3. Three eligible subjects will be enrolled in sequential cohorts at increasing dose levels until at least 1 DLT is observed during the first cycle of vosaroxin therapy. Subjects who receive both doses of vosaroxin will be evaluated for the MTD, DLTs, and safety profile during the first cycle of therapy. Once the MTD has been determined, an expanded evaluation of safety and hematologic response or improvement rate at this dose level will be conducted in additional subjects so that the total number of subjects exposed to this dose level is up to 15 subjects, inclusive of those treated at this dose level in the dose-escalation phase. The exposure of additional subjects at the MTD will provide a better estimate of the toxicity rate. Subjects with a documented response of Complete Response, Partial Response, or hematologic improvement at the end of Cycle 2 may continue to receive vosaroxin for additional cycles at the discretion of the treating investigator and after discussion with the medical staff at Sunesis Pharmaceuticals. There will be a 30-day follow-up period following the termination of study drug treatment.

ELIGIBILITY:
Inclusion Criteria:

* Able to understand and to provide written informed consent
* At least 18 years of age with pathologically confirmed MDS (< 20% blasts in bone marrow, peripheral blood, or both) by WHO classification with an intermediate 2 or high-risk score assessed by IPSS (score ≥ 1.5)
* Must have received at least 4 cycles of decitabine-based or 6 cycles of azacitidine-based therapy and are either refractory to, relapsed after, or are intolerant of prior therapy with either agent.

  1. Primary failure/refractory: Stable or worsening disease after a minimum of 4 cycles of decitabine-based or 6 cycles of azacitidine-based therapy
  2. Secondary failure/relapse: Bone marrow blast count increase or loss of hematologic response after initial treatment response with hypomethylating agent-based therapy
  3. Intolerance: Intolerance of hypomethylating agent-based therapy regardless of number of cycles completed and clinical response
* Eastern Cooperative Oncology Group (ECOG) Performance Status score of 0-2
* Must have a life expectancy of at least 2 months
* Must demonstrate adequate clinical laboratory values (based on local laboratory results) as follows:

  1. Serum creatinine 1.5 ≤ x the upper limit of normal (ULN) or calculated creatinine clearance (CLCR) of ≥ 50 mL/min
  2. Total bilirubin ≤ 1.5 x ULN, higher levels are acceptable if these can be attributed to active hemolysis (as indicated by positive Coomb's test, decreased haptoglobin, Gilbert's disease, elevated indirect bilirubin, and/or lactate dehydrogenase) or ineffective erythropoiesis (as indicated by bone marrow findings).
  3. Aspartate aminotransferase (AST) ≤ 2.5 x ULN
  4. Alanine aminotransferase (ALT) ≤ 2.5 x ULN
  5. Must show adequate cardiac function defined as a left ventricular ejection fraction (LVEF)
* 40% by echocardiogram (ECHO) or multigated acquisition (MUGA) scan
* Must have acceptable recovery from clinically significant non-hematologic toxicity after prior therapy
* Must be infertile or agree to use an effective contraceptive method for the duration of the study and for 30 days after the last dose (for men and women of child-producing potential).

Exclusion Criteria:

* Patients meeting any of the following criteria are excluded:
* Presence of AML (≥ 20% blasts in bone marrow, peripheral blood, or both)
* Presence of serious illness, medical condition, or other medical history, involving the heart, kidney, liver or other organ system, including abnormal laboratory parameters, which, in the opinion of the Investigator, would be likely to interfere with a subject's participation in the study or with the interpretation of the results.
* Have known active central nervous system disease or active, uncontrolled, clinically significant infection(s).
* Have other active malignancies (including other hematologic malignancies) or other malignancies within 12 months before enrollment, except nonmelanoma skin cancer or cervical intraepithelial neoplasia
* Have experienced CTCAE Grade 2 or greater oral mucositis within the last 14 days
* Are receiving any other investigational therapy or protocol-prohibited therapy
* Have received previous treatment with vosaroxin
* Pregnant or breastfeeding females
* Known allergy to D-sorbitol or methanesulfonic acid (excipients used in vosaroxin)
* Treatment with any anticancer therapy (including radiation) within the previous 14 days prior to the first dose of study drug or less than full recovery (CTCAE grade 1) from the clinically significant toxic effects of that treatment.
* Treatment with any investigational drugs within the previous 14 days prior to Cycle 1, Day 1 or ongoing adverse events from previous cancer treatment with investigational drugs, regardless of the time period.
* Have any other medical, psychological, or social condition that, in the opinion of the PI, would contraindicate the patient's participation in the clinical study due to safety or compliance with clinical study procedures

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2013-10-25 (Actual); Primary Completion 2015-01-19 (Actual); Study Completion 2015-01-19 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Gail Roboz, MD, Principal Investigator — Weill Medical College of Cornell University
Locations (1):
- Weill Cornell Medical College, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Vosaroxin: All Patients Receiving Dose Level 1: Vosaroxin 50 m: All patients will receive vosaroxin according to the dose cohort in which they are enrolled.
  Vosaroxin: Dose level 1: Vosaroxin 50 mg/m^2 IV on Days 1 and 4 of 28 day cycle
- Dose Level 2: Vosaroxin 72 mg/m^2 IV on Days 1 and 4 of 28 Day: All patient receiving Dose level 2: Vosaroxin 72 mg/m^2 IV on Days 1 and 4 of 28 day cycle
- Dose Level 3: Vosaroxin 50 mg/m^2 IV on Days 1, 4, 8 and 11 of: All patient receiving Dose level 3: Vosaroxin 50 mg/m^2 IV on Days 1, 4, 8 and 11 of 28 day cycle
Period: Overall Study
Arm/Group | Vosaroxin: All Patients Receiving Dose Level 1: Vosaroxin 50 m | Dose Level 2: Vosaroxin 72 mg/m^2 IV on Days 1 and 4 of 28 Day | Dose Level 3: Vosaroxin 50 mg/m^2 IV on Days 1, 4, 8 and 11 of
Started | 4 | 4 | 2
Completed | 3 | 3 | 2
Not Completed | 1 | 1 | 0
Not completed — Death | 1 | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Dose Level 1: Vosaroxin 50 mg/m^2 IV on Days 1 and 4 of 28 Day: All patients will receive vosaroxin according to the dose cohort in which they are enrolled.
  Vosaroxin: Dose level 1: Vosaroxin 50 mg^m2 IV on Days 1 and 4 of 28 day cycle
- Dose Level 2: Vosaroxin 72 mg/m^2 IV on Days 1 and 4 of 28 Day: All patients will receive vosaroxin according to the dose cohort in which they are enrolled.
  Dose level 2: Vosaroxin 72 mg^m2 IV on Days 1 and 4 of 28 day cycle
- Dose Level 3: Vosaroxin 50mg/m^2 IV on Days 1, 4, 8 and 11 of: All patients will receive vosaroxin according to the dose cohort in which they are enrolled.
  Dose level 3: Vosaroxin 50 mg^m2 IV on Days 1, 4, 8 and 11 of 28 day cycle
- Total: Total of all reporting groups
Arm/Group | Dose Level 1: Vosaroxin 50 mg/m^2 IV on Days 1 and 4 of 28 Day | Dose Level 2: Vosaroxin 72 mg/m^2 IV on Days 1 and 4 of 28 Day | Dose Level 3: Vosaroxin 50mg/m^2 IV on Days 1, 4, 8 and 11 of | Total
Number analyzed (Participants) | 4 | 4 | 2 | 10
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 0 | 0 | 0 | 0
  >=65 years | 4 | 4 | 2 | 10
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 2 | 1 | 4
  Male | 3 | 2 | 1 | 6
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 2 | 2 | 1 | 5
  Unknown or not reported | 2 | 2 | 1 | 5
Region of Enrollment [Number; unit: participants]
  United States | 4 | 4 | 2 | 10

OUTCOME MEASURES:

1. Primary Outcome: Dosage Determination for IV-infusion of Vosaroxin in Int-2 or High-risk Mds
Description: Maximum tolerated dose of vosaroxin for short IV infusion in INT-2 or high-risk MDS
Time Frame: 1 year
Population: All participants who received at least one dose of Vosaroxin were assessed for DLT in the first cycle of therapy. For this study. MTD is defined as the highest dose level at which no more than 33% of the patients observed at a given dose level experience a DLT.
Measure: Number; unit: mg/m^2
Groups:
- All Study Participants: All patients will receive vosaroxin according to the dose cohort in which they are enrolled.
  Dose level 1: Vosaroxin 50 mg/m^2 IV on Days 1 and 4 of 28 day cycle Dose level 2: Vosaroxin 72 mg/m^2 IV on Days 1 and 4 of 28 day cycle Dose level 3: Vosaroxin 50 mg/m^2 IV on Days 1, 4, 8 and 11 of 28 day cycle
Arm/Group | All Study Participants
Number analyzed (Participants) | 10
mg/m^2 | 200

2. Secondary Outcome: Number of Subjects Who Experience a Response
Description: Evaluate the clinical activity of vosaroxin in MDS subjects by observing number of patients who achieve complete remission.
Time Frame: 15 months
Measure: Count of Participants; unit: Participants
Groups:
- Vosaroxin: Dose Level 1: Vosaroxin 50 mg/m^2 IV on Days 1 & 4: All patients will receive vosaroxin according to the dose cohort in which they are enrolled.
  Vosaroxin: Dose level 1: Vosaroxin 50 mg/m^2 IV on Days 1 and 4 of 28 day cycle
- Dose Level 2: Vosaroxin 72 mg/m^2 IV on Days 1 and 4 of 28 Day: Dose level 2: Vosaroxin 72 mg/m^2 IV on Days 1 and 4 of 28 day cycle
- Dose Level 3: Vosaroxin 50 mg/m^2 IV on Days 1, 4, 8 and 11 of: Dose level 3: Vosaroxin 50 mg/m^2 IV on Days 1, 4, 8 and 11 of 28 day cycle
Arm/Group | Vosaroxin: Dose Level 1: Vosaroxin 50 mg/m^2 IV on Days 1 & 4 | Dose Level 2: Vosaroxin 72 mg/m^2 IV on Days 1 and 4 of 28 Day | Dose Level 3: Vosaroxin 50 mg/m^2 IV on Days 1, 4, 8 and 11 of
Number analyzed (Participants) | 4 | 4 | 2
Participants | 0 | 0 | 0

3. Secondary Outcome: Number of Transfusions Required During Treatment With Vosaroxin
Description: Characterize the blood product transfusion requirements in this patient population when treated with vosaroxin
Time Frame: 15 months
Measure: Mean (Full Range); unit: Transfusions
Groups:
- Vosaroxin: Dose Level 1: Vosaroxin 50 mg^m2 IV on Days 1 and 4: All patients will receive vosaroxin according to the dose cohort in which they are enrolled.
  Vosaroxin: Dose level 1: Vosaroxin 50 mg^m2 IV on Days 1 and 4 of 28 day cycle
- Dose Level 2: Vosaroxin 72 mg^m2 IV on Days 1 and 4 of 28 Day: Dose level 2: Vosaroxin 72 mg^m2 IV on Days 1 and 4 of 28 day cycle
- Dose Level 3: Vosaroxin 50 mg^m2 IV on Days 1, 4, 8 and 11 of: Dose level 3: Vosaroxin 50 mg^m2 IV on Days 1, 4, 8 and 11 of 28 day cycle
Arm/Group | Vosaroxin: Dose Level 1: Vosaroxin 50 mg^m2 IV on Days 1 and 4 | Dose Level 2: Vosaroxin 72 mg^m2 IV on Days 1 and 4 of 28 Day | Dose Level 3: Vosaroxin 50 mg^m2 IV on Days 1, 4, 8 and 11 of
Number analyzed (Participants) | 4 | 4 | 2
Transfusions | 19.8 [2 to 44] | 22.5 [12 to 33] | 22 [17 to 27]

ADVERSE EVENTS:
Time Frame: Adverse events were collected over a period of 15 months.
Description: The adverse events and SAEs were assessed and graded by the principal investigator throughout the study.
Groups:
- Dose Level 1: Vosaroxin 50 mg/m2 IV on Days 1 and 4 of 28 Day: Vosaroxin: Dose level 1: Vosaroxin 50 mg/m2 IV on Days 1 and 4 of 28 day cycle
- Dose Level 2: Vosaroxin 72 mg/m2 IV on Days 1 and 4 of 28 Day: Dose level 2: Vosaroxin 72 mg/m2 IV on Days 1 and 4 of 28 day cycle
- Dose Level 3: Vosaroxin 50 mg/m2 IV on Days 1, 4, 8 and 11 of: Dose level 3: Vosaroxin 50 mg/m2 IV on Days 1, 4, 8 and 11 of 28 day cycle
Arm/Group | Dose Level 1: Vosaroxin 50 mg/m2 IV on Days 1 and 4 of 28 Day | Dose Level 2: Vosaroxin 72 mg/m2 IV on Days 1 and 4 of 28 Day | Dose Level 3: Vosaroxin 50 mg/m2 IV on Days 1, 4, 8 and 11 of
All-Cause Mortality (participants affected / at risk) | 1/4 | 1/4 | 0/2
Serious Adverse Events (participants affected / at risk) | 3/4 | 1/4 | 2/2
Other Adverse Events (participants affected / at risk) | 3/4 | 3/4 | 2/2
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Dose Level 1: Vosaroxin 50 mg/m2 IV on Days 1 and 4 of 28 Day (N=4) | Dose Level 2: Vosaroxin 72 mg/m2 IV on Days 1 and 4 of 28 Day (N=4) | Dose Level 3: Vosaroxin 50 mg/m2 IV on Days 1, 4, 8 and 11 of (N=2)
Febrile Neutropenia (Blood and lymphatic system disorders) | 3 | 0 | 1
Non- Cardiogenic Shock (General disorders) | 0 | 1 | 0
Sudden Death (General disorders) | 1 | 0 | 0
Respiratory Distress (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Disease Progression (Blood and lymphatic system disorders) | 0 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Dose Level 1: Vosaroxin 50 mg/m2 IV on Days 1 and 4 of 28 Day (N=4) | Dose Level 2: Vosaroxin 72 mg/m2 IV on Days 1 and 4 of 28 Day (N=4) | Dose Level 3: Vosaroxin 50 mg/m2 IV on Days 1, 4, 8 and 11 of (N=2)
Diarrhea (Gastrointestinal disorders) | 2 | 2 | 2
Fatigue (General disorders) | 3 | 1 | 1
Febrile Neutropenia (Blood and lymphatic system disorders) | 3 | 1 | 1
Constipation (Gastrointestinal disorders) | 3 | 1 | 0
Oral Thrush (Infections and infestations) | 1 | 1 | 0
Epistaxis (General disorders) | 2 | 1 | 1
Nausea (Gastrointestinal disorders) | 2 | 3 | 1
Vomiting (Gastrointestinal disorders) | 1 | 2 | 0
Mucositis (Gastrointestinal disorders) | 1 | 1 | 2
Bacterimia (Infections and infestations) | 0 | 1 | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No